CLINICAL TRIAL: NCT03703804
Title: The AfterBabyBodyStudy- Testing Manual Examination Methods and Exercise Effects on Muscular Recovery After Pregnancy
Brief Title: AfterBabyBodyStudy- Testing Manual Examination Methods and Exercise Effects on Muscular Recovery After Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Maria Larsson, Associate Professor, Vastra Gotaland Region
Other Study IDs: VGFOUREG-832541
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Postpartum Period; Pelvic Floor; Diastasis Recti; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women postpartum: Women -over 18 years, ability to understand Swedish in spoken and written terms, gave birth to a child approximately 3 months ago via vaginal delivery or cesarean section will be included. Exclusion criteria will be chronic pain in the pelvis or back (defined as pain in pelvic or back in more than 3 months before pregnancy), major rupture of the pelvic floor at delivery e.g. sphincter rupture grade III/IV or other diseases or surgery that prevents examination of the pelvic floor or abdominal muscles.

SUMMARY:
Exercising postpartum is important for the health of mother and child. However, there are physical changes postpartum which can prevent women from exercising postpartum. About 30% of women postpartum have problems with stress urinary incontinence. Almost as many have a remaining separation of the two parts of the muscle rectus abdominis. Over the last decenium there has been an increased interest but also disparate information about these conditions. This has led to an increased uncertainty among women who wants to resume exercising postpartum. More and more women seek help of physiotherapists to verify an appropriate function in their muscles after pregnancy. However, reliable and valid examination methods are scarce and it is unclear how to interpret the examination results to give individualized exercise advice.

The aim of this study is to test the reliability of examination methods for the pelvic floor function and separation of the rectus abdominis and the criterion validity of these examination methods regarding exercising without leaking urine and lumbopelvic pain. Another aim is to identify if exercising postpartum has effects on the function of the muscles and (less) leaking of urine and lumbopelvic pain/disability.

Recruitment of 300 women approximately 8 weeks postpartum in the Region Västra Götaland. For testing interrater reliability on manual examination of the pelvic floor and the separation of the rectus abdominis by caliper two physiotherapists will examine the participants´ pelvic floor and abdominal muscles. The examinations will be tested for criterion validity using a questionnaire for pelvic floor function, lumbopelvic pain/disability and physical activity level. In an observational component of this study the questionnaire will also be used to evaluate the effects of exercising postpartum on the recovery of pelvic floor and abdominal muscles at 6, 9 and 12 months postpartum.

This study will provide knowledge about the reliability of examination methods for pelvic floor function and separation of the rectus abdominis, their correlation to urinary leakage and pain/disability (criterion validity) and the effects of exercising on muscle function postpartum.

DETAILED DESCRIPTION:
Introduction Exercising postpartum is important for the health of mother [1-3] and child [4]. However, there are physical changes postpartum which can prevent women from exercising postpartum. About 30% of women postpartum have problems with stress urinary incontinence [5]. Between 20-50% of women describe that urine leakage impact their physical activity level [6-8]. Another concern is a remaining separation of the two parts of the rectus abdominis (diastasis rectus abdominis-DRA) which is present in about 30% of women one year postpartum [9]. There is an ongoing discussion about if the DRA is a cause for instability and it is controversial if a DRA is a source for low back and pelvic pain and pelvic floor dysfunction [9-12]. Discussions about how heavy lifting of the growing child and different exercises can harm or benefit the DRA [13] cause an uncertainty among women who want to exercise postpartum. In recent years an increasing number of women are seeking help from physiotherapists in primary care to get physiotherapeutic examination and advice before resuming exercising.

Physiotherapists assess the pelvic floor and abdominal muscles postpartum. Their standard method for pelvic floor muscles evaluation is vaginal palpation using the modified oxford scale [14, 15]. Vaginal palpation is the only method evaluating the ability to perform a correct contraction described as a squeeze with lift- the pelvic floor function [15]. However, researchers are still struggling to rate this function on a scale. The challenge is to rate two movements in one scale [14, 16]. Current studies often just assess the strength component of the contraction [14, 16] with just fair interrater reliability. Other researchers developed scales assessing different qualities of function [17-19] which makes them difficult to apply clinically while palpating at the same time. In the physiotherapeutic assessment the function of a muscle is important. In this study functional components like in the Devreese [17] or Brink scale [20] will be added to the modified oxford scale. Defining the values of the oxford scale more functionally creates the hypothesis that physiotherapists will have easier to agree in their assessments. Another question is which function in the pelvic floor is requested to resume exercising postpartum without leaking urine. The assumption that a strong pelvic floor leads to less stress urinary incontinence is discussed [21, 22]. However, pelvic floor training shows good effect against urinary incontinence [23], According to our knowledge is the correlation between function and exercising postpartum without leaking urine not investigated yet.

For examination of the DRA 96 % of physiotherapists specialized in women´s health use the finger-width method [9, 13]. This method has weaker interrater reliability than instrumental measurement methods [24] and is inaccurate due to variations of finger-width [25]. Assessment of the DRA with a caliber shows almost equally good accuracy like ultrasound assessment [24, 26], it allows the documentation of changes eg the recovery postpartum. However, below 2 % of physiotherapists are using caliper for assessment of postpartum women [13], the interrater reliability is not tested yet. Furthermore there is no international consensus about how to classify the DRA [24], and it is still discussed which width of the DRA can be associated with a dysfunction such as lumbopelvic pain or stress urinary incontinence [9, 10].

The recovery of the pelvic floor and the abdominal muscles occur under the first year after giving birth [9, 27]. International guidelines for exercise postpartum are still scarce and not based on results of RCT´s; especially when it comes to exercises which put high strain on the pelvic floor [28-30]. If and when exercising affects the recovery of pelvic floor function and DRA postpartum is not yet known [6, 22, 31-35]. There are two different hypothesis regarding effects of physical training on the pelvic floor a) physical training is strengthening or b) physical training is weakening the pelvic floor [22, 36]. If physical training in the early postpartum period leads to a better pelvic floor function and less urinary incontinence needs to be investigated.

The effects of different abdominal exercises on the recovery of the DRA is controversy discussed [34, 37, 38]. A review based on low quality studies suggest that all physical activity improves the DRA postpartum [34]. Little is known about the effects of different types of exercising on the recovery of the DRA and further research is needed [39, 40].

The general aim The overall purpose of this thesis is to investigate physiotherapeutic examination methods postpartum and evaluate the effects of exercising in the recovery of pelvic floor function and DRA postpartum.

Clinical implication:

The knowledge gained from this thesis will help to improve our physiotherapeutic examination methods postpartum and be able to give more evidence based exercise advice for a safe resumption of an active lifestyle postpartum.

Included studies This trial will include two studies: 1) a reliability and validity study of examination methods, 2) an observational study. Both studies will use the same recruitment process: Women will be invited to participate via posters at the Swedish antenatal centers in the Region Västra Götaland and social media. Women -over 18 years, ability to understand Swedish in spoken and written terms, gave birth to a child approximately 3 months ago via vaginal delivery or cesarean section will be included. Exclusion criteria will be chronic pain in the pelvis or back (defined as pain in pelvic or back in more than 3 months before pregnancy), major rupture of the pelvic floor at delivery e.g. sphincter rupture grade III/IV or other diseases or surgery that prevents examination of the pelvic floor or abdominal muscles.

Study 1 Interrater reliability and criterion validity of physiotherapeutic examination methods of pelvic floor and DRA postpartum Aims: To evaluate the reliability of examination methods for the pelvic floor and DRA. To test the criterion validity of these two examination methods against the ability to exercise without/less leaking urine or experiencing lumbopelvic pain/ disability.

Method:

The data will be collected via manual examination and a questionnaire. The manual examinations will take place at baseline (approximately 9-12 weeks postpartum) and at three follow-ups.

To evaluate the interrater reliability of manual examination methods for the pelvic floor function and the DRA, the participants receive a physiotherapeutic examination of their pelvic floor and DRA at baseline. The same examination will be conducted by the two physiotherapists in random order with a half hour break in between, the two physiotherapists will be blinded to each other's assessments. They will follow a standardized protocol .

A questionnaire will be used after the manual examination to test the criterion validity of the manual examination methods and the ability to exercise without leaking urine or experiencing lumbopelvic pain/disability. The questionnaire includes 1) the ICIQ-UI Short Form which is brief questionnaire to assess the impact of symptoms of incontinence on quality of life, fully validated and available in Swedish [41] 2) The Oswestry disability index measures the subjective level of function (disability) in daily activities in patients with low back pain [42] 3) The Pelvic Girdle Questionnaire (PGQ) which is a self-reported questionnaire and has high test-retest reliability and good construct validity to test pelvic girdle pain in pregnancy and the postpartum period [43]. The respondents report if and which type of physical activity/training cause them to experience urine loss [8]. The results of the questionnaires will be tested against the results of the manual examinations.

After the first examination at baseline the participants will be manually examined by one of the physiotherapists and fill out the above-described questionnaire in a three months interval (approximately at 6, 9 and 12 months postpartum).

The data will be analyzed using the program IBM SPSS Statistics 22. For interrater reliability a kappa-test will be used to analyze the consistency between the results of manual examination of the two physiotherapists. In this study, the degree of consistency between the two investigators is determined by Kappa value and standard error for manual examination. In addition the Svensson method will be used [44]. For testing the criterion validity of the manual examinations and the ability to exercise without/less leaking urine or experiencing lumbopelvic pain/disability a Svensson MA and Gamma correlation will be used. Associations between pelvic floor function and DRA and urinary leakage and pain/disability measured via instruments (ICIQ-UI short form, Oswestry Disability Index and PGQ, physical activity causing leakage) will be calculated. Criterion validity will be calculated for the first examination at baseline, 6, 9 and 12 months postpartum in order to spread the different variables e g pelvic floor strength/DRA can be expected to be weak/separated at first, but higher at last measurement, as well as urine leakage/pain/disability.

Study 2:

Exercise behavior of postpartum women postpartum and its effects on the pelvic floor and abdominal muscle function.

Aims: To investigate whether early return to exercise postpartum and/or specific types of exercises postpartum (high/low impact aerobics training, strenuous training) affects the recovery of pelvic floor function and DRA.

Method: All data will be collected by the manual examinations (baseline, 6, 9 and 12 months postpartum), the above-described questionnaire which includes for this part of the thesis, two self-reported leisure -time questionnaires: 1) assessing the frequency of 14 different exercises in the last month [45] and 2) assessing the physical activity level according to the public health recommendation of the American college of Sport´s medicine (ACSM) and American Heart Association (AHA) [46] and questions about age, weight and length (BMI), further pregnancies, delivery modes, perineal tear and breastfeeding.

Changes in the pelvic floor function and DRA at the manual examination from baseline to 6, 9 and 12 months postpartum will be compared between the groups "early returned to exercising" and "not returned to exercising" via Wilcoxon rank test. For this study "early return to exercising" is defined as exercising more than strolling at baseline reported via questionnaire, and "not returned to exercising" is defined as if the only reported activity is strolling at 9 months postpartum. A linear regressions analysis will be used to control for others parameters which can influence changes of the pelvic floor function and DRA like age, BMI, type of delivery, number of deliveries, type of perineal tear and instrumental delivery (if known) and possible breastfeeding. Type of exercising will be classified in the questionnaire and divided in seven groups[45]. The groups will be compared regarding changes in the pelvic floor function and DRA between the manual examination at baseline and at 9 months postpartum via Kruskal Wallis test. A p-value 0.05 will be considered as statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Women -over 18 years, ability to understand Swedish in spoken and written terms, gave birth to a child approximately 3 months ago via vaginal delivery or cesarean section will be included.

Exclusion Criteria:

* chronic pain in the pelvis or back (defined as pain in pelvic or back in more than 3 months before pregnancy),
* major rupture of the pelvic floor at delivery e.g. sphincter rupture grade III/IV
* other diseases or surgery that prevents examination of the pelvic floor or abdominal muscles.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women over 18 years old, gave birth via vaginal delivery or c-section
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor function | From baseline to 12 month follow upp
  Pelvic floor function will be rated on a modified oxford scale (0 = no contraction, 1 = flicker, 2 = weak, no lift, 3 = good contraction with lift, 4 = maximal contraction (with lift) and 5 = maximal contraction with lift over 5 seconds.
Diastasis recti abdominis | From baseline to 12 month follow upp
  measured in mm by a caliper
Urinary incontinence | From baseline to 12 month follow upp
  Urinary incontinence assessed by ICIQ-UI short form (rated from 0-21, + questions about functional leakage)
Lumbopelvic pain/disability | From baseline to 12 month follow upp
  assessed by oswestry disability index/Roland morris disability index (0-100% function)/pelvic girdle pain questionnaire (0-100% function)

CONTACTS AND LOCATIONS:
Locations (1):
- Närhälsan Göteborg, Gothenburg, Västra Götalandregionen, Sweden

REFERENCES:
- [Derived] Vesting S, Gutke A, Fagevik Olsen M, Praetorius Bjork M, Rembeck G, Larsson MEH. Can Clinical Postpartum Muscle Assessment Help Predict the Severity of Postpartum Pelvic Girdle Pain? A Prospective Cohort Study. Phys Ther. 2022 Dec 30;103(1):pzac152. doi: 10.1093/ptj/pzac152. PMID 36326139
- [Derived] Vesting S, Olsen MF, Gutke A, Rembeck G, Larsson MEH. Clinical assessment of pelvic floor and abdominal muscles 3 months post partum: an inter-rater reliability study. BMJ Open. 2021 Sep 2;11(9):e049082. doi: 10.1136/bmjopen-2021-049082. PMID 34475166